CLINICAL TRIAL: NCT06624514
Title: Mobile Health Reaction Time and Behavior Study
Brief Title: mHealth Behavior Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00138757
Record Dates: First submitted 2024-09-20; First posted 2024-10-03 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Alcohol Consumption; Condom Use
Keywords: Alcohol; condoms; Sexual Assault; Risky Sex
MeSH Terms: conditions — Alcohol Drinking | interventions — Sensitivity Training Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group (Experimental): This arm receives a version of the AAT used as an Approach Bias Modification (ABM) intervention, to retrain participants' implicit biases toward or away from stimuli by presenting the target stimuli predominantly in one format (e.g., push or pull).
  Interventions: Behavioral: Training Group
- Control (Sham Comparator): No treatment version of the AAT used as an Approach Bias Modification (ABM) intervention will be used in this group.
  Interventions: Behavioral: Sham Training Group

INTERVENTIONS:
Behavioral: Training Group — Implicit approach bias is the behavioral action tendency to be faster to approach rather than avoid cues for a stimulus category. The Approach-Avoidance Task (AAT)is a computerized program in which participants make approach or avoidance movements in response to an irrelevant feature of an image presented on a computer screen (e.g., push when in portrait, pull when in landscape). The intervention in this study is a treatment version of the AAT used as an Approach Bias Modification (ABM) intervention, to retrain participants' implicit biases toward or away from stimuli by presenting the target stimuli predominantly in one format (e.g., push or pull).
  Arms: Training Group
Behavioral: Sham Training Group — A sham-training control condition
  Arms: Control

SUMMARY:
The goal of this clinical trial is to learn if a brief task completed on a smartphone can reduce alcohol use and risky sexual behavior among women between the ages of 18 and 25 who have a history of experiencing sexual assault or an unwanted sexual experience. The main questions it aims to answer are:

* Does the smartphone task change approach biases for alcohol and condom-related images?
* Does the smartphone task reduce alcohol use and risky sexual behavior?

Researchers will compare the smartphone task to a sham control to see if the smartphone task changes biases and behavior.

Participants will:

* Complete a baseline assessment battery of questionnaires
* Complete either the intervention smartphone task or the sham smartphone task on four consecutive days.
* Complete a follow-up assessment one week after finishing the four tasks
* Complete a three-month follow-up

ELIGIBILITY:
Inclusion Criteria:

* Adult women who report lifetime experience sexual assault,
* Consume alcohol at least moderately (e.g., at least seven drinks per week; NIAAA, 2015),
* Have engaged in sexual intercourse with a casual, non-committed male partner without a condom at least three times during the three months prior to data collection.

Exclusion Criteria:

* Active homicidal or suicidal ideation;
* History of or current psychotic disorders as the study protocol may be therapeutically insufficient;
* Previously identified as having a Pervasive Developmental Disability.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Participants will be adult women who:
  * report lifetime experience sexual assault,
  * consume alcohol at least moderately (e.g., at least seven drinks per week; NIAAA, 2015),
  * have engaged in sexual intercourse with a casual, non-committed male partner without a condom at least three times during the three months prior to data collection.
Enrollment: 46 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Approach Bias | 3-months post final intervention session
  At one-week and three-months following the completion of the final study interventional session, participants will complete the AAT Assessment Procedure and complete the baseline questionnaire battery to assess alcohol and condom use since the previous appointment.
Condom Use | Three-Months
  Condom use over the past three months will be measured via the NIDA HIV Risk Measure (HRM).
Alcohol Use | Three-Months
  Alcohol use will be assessed at a three-month follow-up using the Daily Drinking Questionnaire - Revised (DDQ-R).

CONTACTS AND LOCATIONS:
Overall Officials: Austin Hahn, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (1):
  • Informed Consent Form (2025-01-21): https://cdn.clinicaltrials.gov/large-docs/14/NCT06624514/ICF_001.pdf